CLINICAL TRIAL: NCT01979419
Title: Korea Alzheimer's Disease Neuroimaging Initiative
Acronym: K-ADNI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Korean Alzheimers' Disease Neuroimaing Intitiative (Other)
Responsible Party: Principal Investigator, Seong Yoon Kim, MD, PhD, Professor, Department of Psychiatry, Asan Medical Center, Korean Alzheimers' Disease Neuroimaing Intitiative
Other Study IDs: HI12C0713
Record Dates: First submitted 2013-10-21; First posted 2013-11-08 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease; Subcortical Vascular Dementia
Keywords: mild cognitive impairment; Alzheimer's disease; subcortical Vascular Dementia; amyloid; plaques; neuroimaging; biomarkers; cognition disorder; early detection; pre-dementia; dementia; vascular MCI
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular; Plaque, Amyloid; Cognition Disorders; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Blood, Serum, CSF
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- cognitively normal: MRI scans, PET scans, lumbar puncture
- mild cognitive impairment: MRI scans, PET scans, lumbar puncture
- Alzheimer's Disease: MRI scans, PET scans, lumbar puncture
- vascular MCI: MRI scans, PET scans, lumbar puncture
- subcortical ischemic vascular dementia: MRI scans, PET scans, lumbar puncture

SUMMARY:
PRIMARY OBJECTIVES

-Establish a registry for Alzheimer's disease (AD) and subcortical ischemic vascular dementia (SIVD)

STUDY DESIGN

-This is a non-randomized, natural history, observational, registry study.

SAMPLE SIZE AND RECRUITMENT

- Five hundred subjects will be enrolled at each clinical site (50 NC, 200 with MCI, 50 with AD, 100 with vMCI, and 100 with SIVD)

SUMMARY OF KEY ELIGIBILITY CRITERIA

* Newly enrolled subjects will be between 50-80 (inclusive) years of age.
* 1) Cognitively Normal Subjects
* 2) MCI subjects
* 3) AD subjects
* 4) vMCI or SIVD

PROCEDURES

* Recruited subjects will have clinical/cognitive assessments, biomarker and genetic sample collection, and imaging.
* Subjects will be followed up for 36 months from the baseline visit. All assessments are to be performed every year from baseline(0, 12, 24, 36 months), except; 1) FDG-PET and amyloid-PET will be performed every two years, i.e., on baseline and at 24 month visit. 2) CSF collection will also be performed on baseline and at 24 months visit. 3) Clinical/cognitive assessment and MRI evaluation will additionally be done at 6 months from baseline to determine short term change.

OUTCOME MEASURES

* Group differences for each clinical, cognitive, biochemical, and imaging measurement.
* Rate of conversion or change of disease severity will be evaluated among all groups
* Correlations among biomarkers and biomarker changes

DETAILED DESCRIPTION:
The major goals of K-ADNI are to:

1. Establish a registry for Alzheimer's disease (AD) and subcortical ischemic vascular dementia (SIVD)

   * Collect longitudinal clinical, imaging, genetic, and biochemical biomarker data for clinical and neuroscience studies on 500 subjects in five diagnostic categories: cognitively normal control (NC), mild cognitive impairment (MCI), mild AD, vascular MCI (vMCI), and SIVD.
   * The following measurements known as representative parameters of dementia progress will be included. 1) clinical characteristics, 2) neuropsychological test, 3) structural and functional magnetic resonance image (MRI), 4) Fludeoxyglucose (FDG)-positron emission tomography (PET), 5) amyloid PET (18F-flutemetamol), 6) cerebrospinal fluid (CSF) and blood sample, 7) genetic analysis.
2. Determination of factors that are crucial in the aggravation or deterrence of progress of dementia syndrome, so that these factors can be used as predictors and outcome measures of AD and SIVD

   * Determine the relationships among clinical, imaging, genetic, and biochemical biomarker characteristics of the entire spectrum of AD, as the pathology evolves from normal aging through very mild symptoms, to MCI, and finally to dementia.
   * Also, determine the relationship among clinical, imaging, genetic, and biochemical biomarker characteristics of the vascular MCI (vMCI) and SIVD, which is an important sub-population of dementia syndrome especially in Asian population.
3. Identification of surrogate markers for new drug development in patients with AD and SIVD

   - Identify prognostic markers of AD and SIVD, identify outcome measures that can be used in clinical trials, and help develop the most effective clinical trial scenarios for new drugs.
4. Development of the standard model for acquiring multi-site neuroimaging study data - Develop improved methods which will lead to uniform standards for acquiring longitudinal multi-site clinical, MRI, PET, and other biological markers (blood, CSF, gene) data on patients with AD, MCI, vMCI, SIVD, and elderly controls.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitively Normal Subjects

   * Mini-Mental State Examination (MMSE) scores between 24-30 (inclusive)
   * Clinical Dementia Rating (CDR)=0
   * non-depressed (Geriatric Depression Scale scores less than 4)
   * no evidence of cognitive impairment
2. MCI subjects

   * MMSE scores between 24-30 (inclusive)
   * a subjective memory concern reported by subject, informant, or clinician
   * objective memory loss measured by age and education year adjusted scores on logical memory sub-test (below -1.5 SD)
   * CDR=0.5
   * preserved activities of daily living, and an absence of dementia.
3. AD subjects

   * MMSE scores between 20-26 (inclusive)
   * CDR= 0.5 or 1.0.
   * meets National Institute of Neurological and Communicative Disorders and Stroke / Alzheimer's Disease and Related Disorders Associations (NINCDS/ADRDA) criteria for probable AD
4. vMCI or SIVD

   * For diagnosis of vMCI or SIVD, it is necessary to meet the above clinical/cognitive test scores of MCI or AD.
   * Presence of vascularity are determined by; 1) more than 2 vascular risk factors in recent 5 years (hypertension, diabetes, stroke, dyslipidemia, other cardiovascular disease, obesity, lack of exercise, and smoking) AND 2) more than 1 evidence of vascular neurological symptom, sign, or history AND 3) neuroimaging evidence of white matter hyperintensity, which is rated moderate or severe on MR T2-weighted image(T2WI) or FLAIR images.

Exclusion Criteria:

* Screening/baseline MRI scan with evidence of infection, infarction, or other focal lesions; Participants with multiple lacunes or lacunes in a critical memory structure are excluded
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body
* Major depression, bipolar disorder as described in Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) within the past 1 year
* Currently treated with medication for obsessive-compulsive disorder or attention deficit disorder
* History of schizophrenia
* History of alcohol or substance abuse or dependence within the past 2 years
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol
* Any significant neurologic disease such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-11; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Rate of dementia conversion or disease severity worsening, evaluated by neuropsychological, MRI, PET, biomarker indices. | 0 Months (Baseline), 6 Mos, 12 Mos, 24 Mos, 36 Mos
  - The rate of decline as measured by clinical dementia rating (CDR) Sum of Boxes

SECONDARY OUTCOMES:
Change from baseline in cognitive, neuroimaging, and biomarker assessments | 0 Months (baseline), 6 Mos, 12 Mos, 24 Mos, 36 Mos
  * The rate of decline as measured by cognitive tests, Activities of Daily Living
  * The rate of volume change of the whole brain, hippocampus, and other structural MRI measures
  * Rates of change of glucose metabolism (FDG-PET)
  * Extent of amyloid deposition as measured by 18F-flutemetamol
  * Correlations among biomarkers and biomarker changes
  * Group differences for each imaging and biomarker measurement

CONTACTS AND LOCATIONS:
Overall Officials: Seong Yoon Kim, MD, PhD, Principal Investigator — Asan Medical Center, Univ. of Ulsan, Medical College
Locations (1):
- Seong Yoon Kim, Seoul, South Korea